CLINICAL TRIAL: NCT02891356
Title: Bone Mass Changes in Anorexia Nervosa Patient Followed During 4 Years and Relationship Between Bone Loss and Adipokines.
Brief Title: Bone Mass Changes in Anorexia Nervosa Patient Followed During 4 Years
Acronym: AMOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_38; 2012-A01009-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa; Osteoporosis
Keywords: Adiponectin; Bone remodelling markers
MeSH Terms: conditions — Anorexia Nervosa; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anorexia patient: Dual Energy X-ray Absorptiometry (DEXA)
  Interventions: Device: DEXA

INTERVENTIONS:
Device: DEXA — The Dual Energy X-ray Absorptiometry (DEXA) is a third generation multi-captor DEXA device that allow short duration measurements. It measures Bone Mineral Density (BMD) at the spine and the femoral neck

SUMMARY:
The mechanism of bone loss in anorexia nervosa is complex. Marrow adipose tissue seems to play a role in the regulation of bone metabolism. Adipocytes secrete cytokines and adipokines that either stimulate or inhibit adjacent osteoblasts. This study consist to explore the relationship in anorexia nervosa patients with change in bone mineral density and adipokines like leptin, adiponectin and Préf-1 Bone mineral densities will be measure in 180 anorexia nervosa patients at inclusion and every two years during 6 years.It is assessed blood and urinary calcium and phosphate levels, bone remodelling markers and adipokines (leptin, adiponectin and Préf-1)

ELIGIBILITY:
Inclusion Criteria:

* anorexia patient defined by DSM IV diagnostic criteria

Exclusion Criteria:

* patient with other psychiatric disease
* patient with other a metabolic bone disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Anorexia patient recruted in psychiatric unit ( hospitalisation and consultation visit)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density by Dual Energy X-ray Absorptiometry (DEXA) | 4 years
  measured the evolution of the bone mineral density in 180 anorexia nervosa patients and the relationship with this change and adipokine

SECONDARY OUTCOMES:
Incidence of osteoporotic fractures | at 2,4 and 6 years
Adiponectin plasma concentration by ELISA | at 2,4 and 6 years
  measurement of circulating biological factors predicative of changes in BMD
Interleukin-7 plasma concentration by ELISA | at 2,4 and 6 years
  measurement of circulating biological factors predicative of changes in BMD

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LEGROUX, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No